CLINICAL TRIAL: NCT05097027
Title: Effects of Blood Flow Restriction on Post-competition Recovery on Semi-professional and Youth Soccer Players
Brief Title: Blood Flow Restriction and Recovery in Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 221CER21
Record Dates: First submitted 2021-10-05; First posted 2021-10-27 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Resistance Training; Recovery
Keywords: Soccer; Blood Flow Restriction; Performance; Active recovery

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood flow restriction recovery (Experimental I) (Experimental): Active recovery program with blood flow restriction using a periodization methodology in soccer. (Post-match +1 training).
  Interventions: Device: Blood flow restriction recovery
- Non-Blood flow restriction recovery (Experimental II) (Experimental): Active recovery program without blood flow restriction using a periodization methodology in soccer. (Post-match +1 training).
  Interventions: Other: Active recovery

INTERVENTIONS:
Device: Blood flow restriction recovery — Soccer players included in experimental group I will carry out this program for 1 week setting the blood pressure to ~ 60% of limb occlusion pressure (LOP). After a month they will carry out the program without restriction of blood flow. Which will consist of a warm-up part with continuous running (5 min), 6 sprints from box to box of the field at 60-70% of a maximum repetition, and an activation part in the form of rounds with the ball.
  Arms: Blood flow restriction recovery (Experimental I)
Other: Active recovery — Soccer players included in experimental group II will carry out this program for 1 week. After a month they will carry out the program with blood flow restriction. Which will consist of a warm-up part with continuous running (5 min), 6 sprints from box to box of the field at 60-70% of a maximum repetition, and an activation part in the form of rounds with the ball.
  Arms: Non-Blood flow restriction recovery (Experimental II)

SUMMARY:
The objective is to evaluate the effects of blood flow restriction training on the post-competition recovery of professional and semi-professional soccer players. Randomized crossover clinical trial, with two intervention groups: Experimental group I will carry out a recovery training based on the use of the blood flow restriction (BFR) on day 1 post-competition. On the other hand, the Experimental II group will perform the same recovery training without the use of BFR. After 1 month the groups will cross their intervention and make the recovery with the opposite method to the initial one. The study will be carried out during the 2021-2022 season, from first regional to third division of Spanish soccer, with soccer teams from the Mallorca Island. Before the competition, the countermovement jump (CMJ) will be evaluated and repeated at 0, 24, and 72 h after the competition. The levels of muscle soreness (DOMS) will be evaluated pre-post-competition 0, 24, 48 and 72h later. The same procedure will be carried out to evaluate muscle fatigue, sleep quality, and stress through a questionnaire that athletes will fill out pre, 0, 24, 48 and 72h after the game. Sociodemographic and anthropometric data will be collected before starting the study.

DETAILED DESCRIPTION:
W-UP:

The warm-up will consist of 5 minutes running slow, 5 minutes mobility, and 5 minutes of running exercises. In addition, the warm-up will contain a familiarization with the jump test.

ELIGIBILITY:
Inclusion Criteria:

* 50 Minutes or more playing during the last match.

Exclusion Criteria:

* No injuries players.

Ages: 14 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Countermovement Jump (CMJ) | Change from Baseline in countermovement Jump (CMJ Test) at 0 hours, 24 hours, 72 hours and 4 weeks
  CMJ Test measured by Force Platform (Vald Performance, Brisbane, QLD)

SECONDARY OUTCOMES:
Change from Baseline in Rating of Perceived Exertion (RPE) | Change from Baseline in RPE at 0 hours, 24 hours, 48 hours, 72 hours and 4 weeks
  Rating of Perceived Exertion (RPE) measured by Borg scale (0=Rest; 1=Really easy; 2=easy; 3=moderate; 4=sort of hard; 5=hard; 6=hard; 7=Really hard; 8= Really hard; 9= Really, really, hard; 10= Maximal)
Change from Baseline in Fatigue | Change from Baseline in Fatigue at 0 hours, 24 hours, 48 hours, 72 hours and 4 weeks
  Fatigue measured by a Wellness Questionary (1= Always tired; 2=More tired than normal; 3=Normal; 4= Fresh; 5= Very fresh)
Change from Baseline in Muscle Soreness | Change from Baseline in Muscle Soreness at 0 hours, 24 hours, 48 hours, 72 hours and 4 weeks
  Muscle Soreness measured by a Wellness Questionary (1=Very sore; 2= Increase in soreness/ tightness; 3=Normal; 4=Feeling good; 5=Feeling great)
Change from Baseline in Sleep Quality | Change from Baseline in Sleep Quality at 0 hours, 24 hours, 48 hours, 72 hours and 4 weeks
  Sleep Quality measured by a Wellness Questionary (1=Insomnia; 2=Restless sleep; 3=Difficulty falling asleep; 4=good; 5=Very restful)
Change from Baseline in Stress | Change from Baseline in Stress at 0 hours, 24 hours, 48 hours, 72 hours and 4 weeks
  Stress measured by a Wellness Questionary (1=Highly stressed; 2=Feeling stressed; 3=Normal; 4=Relaxed; 5=Very relaxed)
Change from Baseline in Mood | Change from Baseline in Stress at 0 hours, 24 hours, 48 hours, 72 hours and 4 weeks
  Mood measured by a Wellness Questionary (1=Highly annoyed / irritable / down; 2=Snappy with team-mates, family and friends; 3=Less interested in others / activities; 4=Generally good mood; 5=Very positive mood)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Castilla López, Principal Investigator — University of Balearic Islands; Natalia Romero Franco, PhD, Study Director — University of Balearic Islands
Locations (1):
- Christian, Palma de Mallorca, Balearic Islands, Spain